CLINICAL TRIAL: NCT03994263
Title: A Pilot and Prospective Study to Observe the Mechanism of Action of Medi-Tate i-Temporary Implantable Nitinol Device (iTind) in Subjects With Symptomatic Benign Prostatic Hyperplasia (BPH) With Magnetic Resonance Imaging (MRI)
Brief Title: A Prospective Study to Observe the Mechanism of Action of the MediTate iTind in Subjects With Symptomatic BPH With MRI
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: low recruitment
Sponsor: Medi-Tate Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MT-09
Record Dates: First submitted 2019-06-18; First posted 2019-06-21 (Actual); Last update posted 2021-10-07 (Actual); Status verified 2021-09

CONDITIONS: BPH

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- iTind arm (Experimental): ITind device implant
  Interventions: Device: ITind device implant

INTERVENTIONS:
Device: ITind device implant — device implanted for 5-7 days

SUMMARY:
A total of up to 15 eligible subjects will be enrolled into this open-labeled one-arm study designed to observe the mechanism of action of iTind when using MRI

DETAILED DESCRIPTION:
Study Objective:

To validate the iTind efficacy by using MRI in subjects with symptomatic BPH. Specifically the pressure points created by the iTind's struts and its implications on blood flow to the prostate will be assessed.

Efficacy Endpoints:

The endpoints of this study are:

* Decrease in transition zone volume
* Monitor size and location of ablative lesions
* Monitor change in time of lesions
* Monitor the correspondence change in prostate tissue All the above will be assessed by using MRI.

ELIGIBILITY:
Inclusion Criteria:

* Subject signed informed consent form (ICF)
* Age 40 and above- Male with symptomatic BPH.
* IPSS symptom severity score ≥ 13
* Peak urinary flow of < 12 ml/sec
* Prostate volume between 25 ml to 80 ml (assessed by pre-operative ultrasound - TRUS)
* Blood CBC and biochemistry up to two weeks before screening, demonstrating: Normal values of the PT, PTT and INR tests (Anticoagulants washout may be done two weeks prior of device implantation)
* Subject able to comply with the study protocol
* Normal urinalysis and negative urine culture
* Subjects that are able to undergo MRI.

Exclusion Criteria:

* A post void residual (PVR) volume > 250 ml measured by ultrasound or acute urinary retention
* Confirmed or suspected bladder cancer;
* Recent (within 3 months) cystolithiasis or hematuria;
* Urethral strictures, bladder neck contracture, urinary bladder stones or other potentially confounding bladder pathology;
* An active urinary tract infection.
* Enrolled in another treatment trial for any disease within the past 30 days.
* Previous colo- rectal surgery (other than hemorrhoidectomy) or history of rectal disease if the therapy may potentially cause injury to sites of previous rectal surgery, e.g., if a transrectal probe is used;
* Previous pelvic irradiation, cryosurgery or radical pelvic surgery;
* Previous prostate surgery, balloon dilatation, stent implantation, laser prostatectomy, hyperthermia, or any other invasive treatment to the prostate
* Median lobe obstruction of the prostate (larger than 1cm).
* Cancer that is not considered cured, except basal cell or squamous cell carcinoma of the skin (cured defined as no evidence of cancer within the past 5 years)
* Patient with renal dysfunction
* Any serious medical condition likely to impede successful completion of the study

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male with symptomatic BPH
Enrollment: 1 (Actual)
Dates: Start 2019-11-18 (Actual); Primary Completion 2021-02-18 (Actual); Study Completion 2021-02-18 (Actual)

PRIMARY OUTCOMES:
AE rate | 12 months
  Incidence (% of subjects) and frequency (no. of events) of device related adverse events.
Unexpected SAE | 12 months
  Incidence (% of subjects) and frequency (no. of events) of unexpected serious adverse events deemed as related to Meditate iTIND and/or to implantation/retrieval procedures.
Device complications | 12 months
  Incidence (% of subjects) and frequency (no. of events) of Meditate iTIND and/or to implantation/retrieval procedures complications

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Bschleipfer, Prof., Principal Investigator — Weiden Clinic
Locations (1):
- Kliniken Nordoberpfalz AG Klinik für Urologie, Kinderurologie und interdisziplinäres Prostatakarzinomzentrum, Weiden, Germany

IPD SHARING:
Plan to Share IPD: No